CLINICAL TRIAL: NCT03227185
Title: Supporting Episodic Memory With Transcranial Direct Current Stimulation in Healthy Young and Elderly Participants as Well as in Individuals With Memory Impairment
Brief Title: Supporting Episodic Memory With Transcranial Direct Current Stimulation in Healthy Controls and Dementia Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients populations included ==> could not be recruited in meaningful numbers to allow conclusions.
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 3351; 2016-02175 (Other: Cantonal Ethics Committee Bern)
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Healthy; Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two possible sequences of stimulation conditions. Group 1 will receive real tDCS stimulation to the left dlPFC during encoding on the first day and sham stimulation on the second day, and group 2 will receive sham stimulation during encoding on the first day and real tDCS on the second day. The participants will be randomized with equal probability to each of the two groups, using block randomization..
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real - sham anodal tDCS (Experimental): Session 1: 20 min of 1 mA anodal tDCS applied via 5x7 cm rubber electrodes over the DLPFC (current density: 0.028 mA/cm2). Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for the duration of the encoding phase.
  Session 2: 30 s of 1 mA anodal tDCS applied via 5x7 cm rubber electrodes over the DLPFC (current density: 0.028 mA/cm2). Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for the duration of the encoding phase.
  Interventions: Device: real anodal transcranial direct current stimulation (tDCS); Device: sham transcranial direct current stimulation (tDCS)
- Sham - real anodal tDCS (Experimental): Session 1: 30 s of 1 mA anodal tDCS applied via 5x7 cm rubber electrodes over the DLPFC (current density: 0.028 mA/cm2). Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for the duration of the encoding phase.
  Session 2: 20 min of 1 mA anodal tDCS applied via 5x7 cm rubber electrodes over the DLPFC (current density: 0.028 mA/cm2). Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for the duration of the encoding phase.
  Interventions: Device: real anodal transcranial direct current stimulation (tDCS); Device: sham transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: real anodal transcranial direct current stimulation (tDCS) — The MR-compatible neuroConn DC-Stimulator MR (neuroCare Group, Ilmenau, Germany) will be used in the study.
Device: sham transcranial direct current stimulation (tDCS) — The MR-compatible neuroConn DC-Stimulator MR (neuroCare Group, Ilmenau, Germany) will be used in the study.

SUMMARY:
Previous studies showed that anodal tDCS applied over the dorsolateral prefrontal cortex (DLPFC) improved episodic memory performance, indicating a possible use as an intervention for patients suffering from memory impairments. At the same time, only scant evidence (provided by functional magnetic resonance imaging (fMRI) and magnetic resonance spectroscopy (MRS)) exists regarding the underlying mechanisms, thus hindering a more targeted application.

The present study aims at establishing a connection between the stimulation-induced change in episodic memory performance on the behavioural level and neurophysiological parameters. TDCS effects and the underlying mechanisms will be compared between different study conditions, receiving either real anodal tDCS or sham stimulation over the left dorsolateral prefrontal cortex during an episodic memory task.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Right-handedness
* Non-smokers
* Native German speakers or comparable level of fluency
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Neurological or psychiatric condition (other than diagnosed cognitive impairment)
* Past head injuries
* Magnetizable implants
* History of seizures
* Current or life-time alcohol or drug abuse
* Pregnancy
* Skin diseases

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
Episodic memory performance - learning curve | 0.25 hours
  Number of encoded words during the three consecutive immediate retrievals in the encoding phase
Episodic memory performance - delayed recall 1 | 20 min after encoding phase
  Number of remembered words in the delayed recall after a short delay at the day of the on-site visit
Episodic memory performance - delayed recall 2 | 1 day after on-site visit
  Number of remembered words one day after learning

SECONDARY OUTCOMES:
Neurotransmitter levels | 0.5 hours
  Changes in neurotransmitter levels (gamma-Aminobutyric acid (GABA) and glutamatergic metabolites (Glx) due to tDCS (comparing pre- and post-stimulation measurements in DLPFC)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Klöppel, Prof, Principal Investigator — University Hospital of Old Age Psychiatry and Psychotherapy
Locations (1):
- University Hospital of Old Age Psychiatry and Psychotherapy, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No